CLINICAL TRIAL: NCT06545149
Title: SUPPLEMENTATION WITH FERMENTED AND BALANCED FOOD WITH BETA GLUCAN FAVORS THE INNATE AND ADAPTATIVE RESPONSE OF PATIENTS ADMITTED TO A MEDICAL CLINIC WARD? A RANDOMIZED TRIAL
Brief Title: SUPPLEMENTATION WITH BETA GLUCAN AND ADAPTATIVE RESPONSE.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Kaiser Clinic and Hospital (Other)
Responsible Party: Principal Investigator, FERNANDO SABIA TALLO, Clinical Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 73701723.8.0000.0281
Record Dates: First submitted 2024-07-02; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Clinical Course
MeSH Terms: conditions — Disease Progression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The group will receive the intervention with coconut wheat
  Interventions: Dietary Supplement: BioNutri AR-1,
- BioNutri AR-1 (Experimental): The group will receive the intervention with fermented and nutritionally balanced food
  Interventions: Dietary Supplement: BioNutri AR-1,

INTERVENTIONS:
Dietary Supplement: BioNutri AR-1, — intervention with fermented and nutritionally balanced food twice a day

SUMMARY:
Abstract: Studies demonstrate that the use of nutritional supplements containing beta-glucans stimulates the immune system, modulates inflammatory activity, and promotes so-called immune training. Beta-glucans are prebiotics that stimulate the growth and activity of gastrointestinal microbiota and inhibit pathogen growth. Nutritional intervention is crucial for patients' positive evolution, and providing a supplement with highly bioavailable nutrients can make a difference in their nutritional, metabolic, and immune status. Therefore, the study aims to verify the effectiveness of the innate and adaptive immune response to a nutritionally balanced fermented food, containing oral or enteral beta-glucans, in patients treated at 3 Emergency Care Units in São José do Rio Preto, São Paulo, Brazil. This is a prospective randomized study with a characteristic design involving patients treated in the medical wards of 3 Emergency Care Unit. The following assessments will be conducted: Global Subjective Assessment for adults and Mini Nutritional Assessment for the elderly, Sociodemographic, and Laboratory Evaluation.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the medical clinic ward

Exclusion Criteria:

Patients unable to swallow

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
length of hospital stay | during hospitalization

SECONDARY OUTCOMES:
need for readmission | up to 24 weeks
need for ICU | up to 24 weeks

IPD SHARING:
Plan to Share IPD: No